CLINICAL TRIAL: NCT02212704
Title: Verticality Perception - Dissociating Head and Trunk Contributors in Healthy Human Subjects
Brief Title: Verticality Perception - Multisensory Contribution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: perception_head_roll_zurich
Record Dates: First submitted 2014-08-06; First posted 2014-08-08 (Estimated); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Verticality Perception in Healthy Human Subjects; Individual Contribution of Different Sensory Systems
Keywords: vestibular; proprioception; spatial orientation; bayesian
MeSH Terms: conditions — Orientation, Spatial | interventions — Vestibular Evoked Myogenic Potentials

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vestibular stimulation (Experimental): This is the experimental paradigm applied in all participants
  Interventions: Other: Vestibular stimulation by use of the turntable (static roll-tilt while the head is roll-tilted relative to the trunk); Other: 3D-video-head impulse testing; Other: Vestibular-evoked myogenic potentials (VEMPs)

INTERVENTIONS:
Other: Vestibular stimulation by use of the turntable (static roll-tilt while the head is roll-tilted relative to the trunk)
Other: 3D-video-head impulse testing — Evaluation of semicircular canal function. This intervention is part of the screening to determine suitability for this study
Other: Vestibular-evoked myogenic potentials (VEMPs) — Evaluation of otolith function. This intervention is part of the screening to determine suitability for this study

SUMMARY:
The purpose of this study is to evaluate the relative contribution of head- and trunk-based sensory systems to internal estimates of direction of gravity in healthy human subjects. To implement this assessment experimentally, the investigators will use a motor-driven 3D-turntable and a thermoplastic mask to keep the head in a stable, either roll-tilted (±30°) or aligned with the trunk. The investigators will then obtain measurements of the subjective visual vertical in seven different whole-body roll positions (max. 90° roll-tilt). Analysis will be driven by a state-of-the art Bayesian integration model. The investigators hypothesize that different sensory input signals are combined in a statistically optimal fashion.

ELIGIBILITY:
Inclusion Criteria:

* ages 18-60 years
* informed consent
* absence of exclusion criteria

Exclusion Criteria:

* peripheral-vestibular deficit
* disturbed consciousness
* history of sensory deficits
* visual field deficits
* other neurological or systemic disorder which can cause dementia or cognitive dysfunction
* intake of antidepressants, sedatives, or neuroleptics
* pregnancy, unless excluded by a negative pregnancy test
* known neck pain or status post neck trauma

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Accuracy and precision of SVV adjustments in different head and trunk roll-tilt positions | During the turntable measurement (90 minutes)

SECONDARY OUTCOMES:
relative contribution of head- and trunk-based sensory systems based on Bayesian modelling | while on the turntable (1.5 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Straumann, Prof, MD, Principal Investigator — University Hospital Zurich, Dept. of Neurology
Locations (1):
- University Hospital Zurich, Dept. of Neurology, Zurich, Canton of Zurich, Switzerland